CLINICAL TRIAL: NCT06416137
Title: Dementia in Migrants Living in Italy: Promoting a Diversity-sensitive Clinical Approach and Provision of Care
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Marco Canevelli, Principal Investigator, Istituto Superiore di Sanità
Other Study IDs: GR-2021-12372081
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dementia; Alzheimer Disease
Keywords: dementia; migrants; cross-cultural
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Migrants: A group of 1,500 migrants with cognitive impairment will be enrolled at CCDDs.
  Interventions: Diagnostic Test: Neuropsychological tests
- Natives: A group of 1,500 natives with cognitive impairment will be enrolled at CCDDs.
  Interventions: Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: Neuropsychological tests — Participants will be assessed with neuropsychological tests and will be collected information about their lifestyle, clinical history and sociodemographic status. Special attention will be paid to the presence of modifiable risk factors for dementia (i.e., low education, hearing impairment, traumatic brain injury, excessive alcohol consumption, obesity, smoking, hypertension, depression, physical inactivity, diabetes, and social isolation).

SUMMARY:
The number of older migrants with cognitive impairment and dementia living in Italy and attending national healthcare services is rapidly increasing. There is a need to develop diversity-sensitive policies and practices to include migrants and people with different cultural values in the public health response to dementia.

DETAILED DESCRIPTION:
Based on the gaps and barriers identified by the ImmiDem study (GR-2016-02364975), the present project aims to:

i) Describe the clinical and sociodemographic characteristics of migrants with cognitive disorders living in Italy, their health outcomes, and their access to healthcare resources; ii) develop and disseminate screening and assessment tools allowing the cross-cultural cognitive examination of individuals with a migration background; iii) raise awareness about dementia among culturally diverse people and train healthcare professionals in how to provide culturally competent care and support for migrants with cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Migrant (person who was not born in Italy) attending an Italian CCDD;
* Presence of a cognitive impairment.

Exclusion Criteria:

* A person without any cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All migrants consecutively referred to CCDDs due to cognitive disturbances in one year will be considered.
  The following definition of migrants will be consistently adopted in the project: any person living in Italy but born abroad, regardless of the legal status, the reason for migration, and the length of the stay (source: International Organization for Migration).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Global cognitive functioning | Baseline
  Global cognitive functioning will be assessed through the Rowland Universal Dementia Assessment Scale (RUDAS). This is a short cognitive screening instrument designed to minimise the effects of cultural learning and language diversity on the assessment of baseline cognitive performance. The score ranges from 0 to 30. Higher scores indicate better cognitive functioning.

SECONDARY OUTCOMES:
Frailty | Baseline
  Frailty will be assessed by computing a Frailty Index (FI) focusing on the clinical history of the patient and collecting diverse deficits. Patients with a higher number of deficits will be considered frailer.
Risk factors | Baseline
  Special attention will be paid to the presence of modifiable risk factors for dementia (i.e., low education, hearing impairment, traumatic brain injury, excessive alcohol consumption, obesity, smoking, hypertension, depression, physical inactivity, diabetes, and social isolation). They will be collected and analyzed through a specific questionnaire.

IPD SHARING:
Plan to Share IPD: Yes
A workshop will be organized at the end of the project for disseminating the study results to major stakeholders (e.g., healthcare professionals, representatives of migrant communities, local authorities).
Supporting Information: Study Protocol, SAP
Time Frame: After 36 months by the beginning of the study

REFERENCES:
- See also: The website created during the first part of this project. — http://www.immidem.it/